CLINICAL TRIAL: NCT05603000
Title: A Randomized Controlled Trial of Emotion Focused Family Therapy for Parents of Children With Mental Health Difficulties
Brief Title: Emotion Focused Family Therapy for Parents of Children With Mental Health Difficulties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Kristel Thomassin, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFFT
Record Dates: First submitted 2022-10-13; First posted 2022-11-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Depression; Behavior Problem
Keywords: children; parents; mental health; emotion; psychotherapy; parent-child relationship
MeSH Terms: conditions — Anxiety Disorders; Depression; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial, consisting of an intervention arm (EFFT) and a waitlist control (delayed intervention) arm, which will occur concurrently.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist (delayed intervention) (No Intervention): No treatment will be administered to participants in this arm until after the 4-month follow-up in-lab assessment is completed.
- EFFT intervention (Experimental): Treatment (6-week group Emotion Focused Family Therapy) will be administered to participants in this arm.
  Interventions: Behavioral: Emotion Focused Family Therapy

INTERVENTIONS:
Behavioral: Emotion Focused Family Therapy — The Emotion Focused Family Therapy (EFFT) intervention for this study will be delivered to groups of four to ten parents over six weekly sessions of two hours each. The goal of EFFT is to teach and empower parents to coach their child to process the emotions at the source of their mental health symptoms, to increase their child's adaptive behaviours, and to repair emotional injuries within the parent-child relationship. EFFT also targets parents' own emotional challenges that may prevent them from feeling capable or being able to support their child's treatment.
  Each EFFT session will include introductions, psychoeducation about emotion and psychopathology, introduction of skills, experiential activities (e.g., chair work), open discussion and feedback, and homework activities covering the foci of EFFT: emotion coaching, behaviour coaching, therapeutic apology, and parental emotion blocks.
  Other Names: EFFT
  Arms: EFFT intervention

SUMMARY:
Emotion Focused Family Therapy (EFFT) is a promising intervention that aims to teach parents advanced skills to support their child's development of emotion skills and increase their adaptive behaviours, potentially leading to improvements in their child's psychological functioning and family functioning more broadly.

This randomized controlled trial (RCT; EFFT vs waitlist control) will (1) test the efficacy of a 6-week group EFFT program on parent and child outcomes and (2) examine maintenance of treatment gains up to four months post-intervention.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will test the efficacy of a 6-week Emotion Focused Family Therapy (EFFT) group program on parent and child outcomes, compared to a waitlist control. Families will be randomized to either the EFFT group treatment or a waitlist. The RCT will evaluate changes in parent functioning, child functioning, and parent-child relationship functioning. A 4-month follow-up will test whether any changes from pre-to-post intervention are maintained at 4 months.

The RCT will also test proposed mechanisms of change (parent-child relationship quality, family functioning) and moderators of treatment effectiveness (parental stress).

ELIGIBILITY:
Inclusion Criteria:

* Parent of child aged 7 to 15 years old with anxiety, depression, or behavioural challenges
* Parent of child is willing to participate in intervention
* Parent is living at home with the child

Exclusion Criteria:

* Parent or child not proficient enough in speaking/understanding English to complete measures or EFFT intervention components
* Parent or child with a severe mental health disorder (e.g., active suicidality and psychosis) is not considered suitable for the trial intervention due to the clinical need for immediate intervention
* Parent or child is actively receiving, or due to receive, intensive psychological intervention focused on cognitive and/or behavioural strategies to intervene with emotional or behavioural difficulties
* Parent or child has any disabilities in language, speech or hearing that would interfere with their completion of the EFFT and measures
* Parent or child are allergic to adhesive electrode gel use in some tasks (i.e., sodium chloride)

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in parental psychopathology symptoms at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured through the Kessler Psychological Distress Scale (K10), a 10-item self report measure of psychological symptoms that parents will complete. Parents will rate the extent to which they are affected by various psychopathology symptoms on a five-point Likert scale from 1 (None of the time) to 5 (All of the time), with greater total scores (range = 10-50) indicating more severe psychopathology.
Change in child psychopathology symptoms at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured through the Behavior and Feelings Survey (BFS), a 12-item measure of child psychopathology symptoms to be completed by both parents (parent-report) and children (youth-report). Parents and children will rate items on a five-point Likert scale from 0 (Not a problem) to 4 (A very big problem), with greater scores (Internalizing subscale range = 0-24; Externalizing subscale range = 0-24; Total score range = 0-48) indicating more severe psychopathology.
Change in parental emotion regulation at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured through the Difficulties in Emotion Regulation Scale (DERS), a 36-item self-report measure of emotion regulation difficulties to be completed by parents. Parents will indicate the frequency with which they experience difficulties with emotion regulation on a five-point Likert scale from 1 (Almost never) to 5 (Almost always), with greater total scores (range = 36-180) indicating greater difficulties with emotion regulation.
Change in child emotion regulation at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured through the Negative Emotionality subscale of the Child and Adolescent Dispositions Scale (CADS), a scale of child emotion regulation to be completed by parents (parent-report) and children (youth-report). Parents and children will rate the seven Negative Emotionality items on a four-point Likert scale from 1 (Not at all) to 4 (Very much/very often) with greater scores (range = 7-28) indicating poorer emotion regulation.
Change in parent-child co-regulation at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured by parent-child synchrony of heart rate variability during the completion of two lab tasks together (conflict discussion and puzzle task).
Change in parent-child relationship functioning at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured by having parents and their children participate in two lab tasks together (conflict discussion and puzzle task) and coding for behavioural observations.

SECONDARY OUTCOMES:
Change in parental emotion socialization at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured through the Coping with Children's Negative Emotions Scale (CCNES), a 12-item self-report measure of parental emotion parenting practices in response to children's expression of negative emotion. Responses are divided into six subscales representing six distinct types of parental responses. The responses will be grouped in two overall scores: Supportive (Expressive Encouragement, Problem-Focused, and Emotion-Focused Reactions) and Unsupportive (Punitive, Minimizing, and Distress Reactions) practices. Parents will rate the likelihood that they would respond in these distinct ways on a seven-point Likert scale from 1 (Very unlikely) to 7 (Very likely), with greater overall scores (range = 1-7) indicating greater levels of each type of parental response.
Change in parental emotion blocks at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured through the Caregiver Traps Scale (CTS), a 14-item self-report measure of parental emotional blocks. Parents will rate each item on a seven-point Likert scale ranging from 1 (Not likely) to 7 (Extremely Likely), with higher total scores (range = 14-98) indicating greater levels of parental emotional blocks.
Change in parental self-efficacy at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured through the Me as a Parent Questionnaire (MaaP), a 16-item self-report measure of parental self-efficacy. Parents will rate the degree to which they agree with statements about their feelings of competence in their parent role on a five-point Likert scale from 1 (Strongly disagree) to 5 (Strongly agree), with greater total scores (range = 16-80) indicating greater parental self-efficacy.
Fidelity of EFFT program | Throughout intervention over 6 weeks
  This outcome will be measured via audiorecording of group sessions. Fidelity scores will be calculated based on content fidelity - i.e., The degree to which providers implemented the key EFFT components, including: behaviour coaching, emotion coaching, parental emotion blocks, therapeutic apology.
Change in perceived parental stress at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  Parents' perceived level of stress related to tasks associated with parenting will be assessed via the Parental Stress Scale. The Parental Stress Scale is an 18-item parent-report measure that assesses perceived parental stress (sample item: "Caring for my child(ren) sometimes takes more time and energy than I have to give") while taking into account positive and negative facets of parenting. The three subscales that comprise the measure (positive emotional benefits of parenting, sense of enrichment and personal fulfillment, and negative components of parenting) can be summed to form a composite score. Items are rated on a five-point Likert scale from 1 (Strongly Disagree) to 4 (Strongly Agree) with lower scores (range = 18-90) indicating lower levels of parenting stress.
Parental treatment satisfaction | At 6 weeks
  Parental treatment satisfaction will be assessed using the parent-report of the Parent/Child Satisfaction Scales, a parent-report measure of satisfaction with child-oriented mental health services. The parent-report measure (sample item: "To what extent has our program met your child's needs?") has shown good internal consistency and test-retest reliability in prior samples of parents of clinic-referred children. Items are rated on a four-point Likert scale from 1 (Quite dissatisfied) to 4 (Very satisfied), with greater total scores (range = 8-32) indicative of higher overall treatment satisfaction.
Parent-reported change in familial functioning at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  Parent report of familial functioning will be assessed via the McMaster Family Assessment Device, a 60-item measure of broad family functioning that can be completed by any measure of the family system. The measure has subscales that assess particular facets of family functioning (e.g., affective responsiveness; "we cry openly"), which can be summed to form a composite score. Items are rated on a four-point Likert scale from 1 (Strongly Agree) to 4 (Strongly Disagree). Item responses are summed and divided by the number of items in the measure to compute a total score (range = 1-4), with lower total scores indicating more adaptive family functioning.
Change in physiological arousal at 6 weeks and 4 months | Change at 6 weeks; Change at 4 months
  This outcome will be measured by parent and child skin conductance levels during the completion of two lab tasks together (conflict discussion and puzzle task).

CONTACTS AND LOCATIONS:
Overall Officials: Kristel Thomassin, Ph.D, Principal Investigator — University of Guelph
Locations (1):
- Maplewoods Centre for Family Therapy and Child Psychology, University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Research Council (US) and Institute of Medicine (US) Committee on the Prevention of Mental Disorders and Substance Abuse Among Children, Youth, and Young Adults: Research Advances and Promising Interventions; O'Connell ME, Boat T, Warner KE, editors. Preventing Mental, Emotional, and Behavioral Disorders Among Young People: Progress and Possibilities. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32775/ PMID 20662125
- [Background] Ogundele MO. Behavioural and emotional disorders in childhood: A brief overview for paediatricians. World J Clin Pediatr. 2018 Feb 8;7(1):9-26. doi: 10.5409/wjcp.v7.i1.9. eCollection 2018 Feb 8. PMID 29456928
- [Background] Campbell SB, Shaw DS, Gilliom M. Early externalizing behavior problems: toddlers and preschoolers at risk for later maladjustment. Dev Psychopathol. 2000 Summer;12(3):467-88. doi: 10.1017/s0954579400003114. PMID 11014748
- [Background] Freuchen A, Kjelsberg E, Lundervold AJ, Groholt B. Differences between children and adolescents who commit suicide and their peers: A psychological autopsy of suicide victims compared to accident victims and a community sample. Child Adolesc Psychiatry Ment Health. 2012 Jan 4;6:1. doi: 10.1186/1753-2000-6-1. PMID 22216948
- [Background] Reef J, Diamantopoulou S, van Meurs I, Verhulst FC, van der Ende J. Developmental trajectories of child to adolescent externalizing behavior and adult DSM-IV disorder: results of a 24-year longitudinal study. Soc Psychiatry Psychiatr Epidemiol. 2011 Dec;46(12):1233-41. doi: 10.1007/s00127-010-0297-9. Epub 2010 Oct 10. PMID 20936464
- [Background] Buckholdt KE, Parra GR, Jobe-Shields L. Intergenerational Transmission of Emotion Dysregulation Through Parental Invalidation of Emotions: Implications for Adolescent Internalizing and Externalizing Behaviors. J Child Fam Stud. 2014 Feb 1;23(2):324-332. doi: 10.1007/s10826-013-9768-4. PMID 24855329
- [Background] Cao M, Powers A, Cross D, Bradley B, Jovanovic T. Maternal emotion dysregulation, parenting stress, and child physiological anxiety during dark-enhanced startle. Dev Psychobiol. 2017 Dec;59(8):1021-1030. doi: 10.1002/dev.21574. Epub 2017 Oct 13. PMID 29027660
- [Background] Fabes RA, Leonard SA, Kupanoff K, Martin CL. Parental coping with children's negative emotions: relations with children's emotional and social responding. Child Dev. 2001 May-Jun;72(3):907-20. doi: 10.1111/1467-8624.00323. PMID 11405590
- [Background] Morris AS, Silk JS, Steinberg L, Myers SS, Robinson LR. The Role of the Family Context in the Development of Emotion Regulation. Soc Dev. 2007 May 1;16(2):361-388. doi: 10.1111/j.1467-9507.2007.00389.x. PMID 19756175
- [Background] Ramsden SR, Hubbard JA. Family expressiveness and parental emotion coaching: their role in children's emotion regulation and aggression. J Abnorm Child Psychol. 2002 Dec;30(6):657-67. doi: 10.1023/a:1020819915881. PMID 12481978
- [Background] Granic I, O'Hara A, Pepler D, Lewis MD. A dynamic systems analysis of parent-child changes associated with successful "real-world" interventions for aggressive children. J Abnorm Child Psychol. 2007 Oct;35(5):845-57. doi: 10.1007/s10802-007-9133-4. Epub 2007 Jun 5. PMID 17549621
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Weisz JR, Vaughn-Coaxum RA, Evans SC, Thomassin K, Hersh J, Ng MY, Lau N, Lee EH, Raftery-Helmer JN, Mair P. Efficient Monitoring of Treatment Response during Youth Psychotherapy: The Behavior and Feelings Survey. J Clin Child Adolesc Psychol. 2020 Nov-Dec;49(6):737-751. doi: 10.1080/15374416.2018.1547973. Epub 2019 Jan 18. PMID 30657721
- [Background] Lahey BB, Applegate B, Chronis AM, Jones HA, Williams SH, Loney J, Waldman ID. Psychometric characteristics of a measure of emotional dispositions developed to test a developmental propensity model of conduct disorder. J Clin Child Adolesc Psychol. 2008 Oct;37(4):794-807. doi: 10.1080/15374410802359635. PMID 18991130
- [Background] Foroughe M, Stillar A, Goldstein L, Dolhanty J, Goodcase ET, Lafrance A. Brief Emotion Focused Family Therapy: An Intervention for Parents of Children and Adolescents with Mental Health Issues. J Marital Fam Ther. 2019 Jul;45(3):410-430. doi: 10.1111/jmft.12351. Epub 2018 Aug 13. PMID 30105875
- [Background] Lafrance Robinson A, Dolhanty J, Stillar A, Henderson K, Mayman S. Emotion-Focused Family Therapy for Eating Disorders Across the Lifespan: A Pilot Study of a 2-Day Transdiagnostic Intervention for Parents. Clin Psychol Psychother. 2016 Jan-Feb;23(1):14-23. doi: 10.1002/cpp.1933. Epub 2014 Nov 23. PMID 25418635
- [Background] Lafrance A, Strahan EJ, Stillar A. Treatment-engagement fears in family-oriented interventions: validation of the caregiver traps scale for eating disorders. Eat Disord. 2022 Nov-Dec;30(6):670-685. doi: 10.1080/10640266.2021.1993706. Epub 2021 Nov 7. PMID 34743672
- [Background] Lafrance A, Henderson KA, Mayman S. Emotion-focused family therapy: A transdiagnostic model for caregiver-focused interventions. American Psychological Association; 2020.
- [Background] Vrana G, Greenberg L. Overview of emotion-focused therapy. In Emotion Focused Family Therapy with Children and Caregivers 2018 Mar 15 (pp. 1-22). Routledge.
- [Background] Strahan EJ, Stillar A, Files N, Nash P, Scarborough J, Connors L, Gusella J, Henderson K, Mayman S, Marchand P, Orr ES. Increasing parental self-efficacy with emotion-focused family therapy for eating disorders: A process model. Person-Centered & Experiential Psychotherapies. 2017 Jul 3;16(3):256-69.
- [Background] Wilhelmsen-Langeland A, Aardal H, Hjelmseth V, Fyhn KH, Stige SH. An emotion focused family therapy workshop for parents with children 6-12 years increased parental self-efficacy. Emotional and Behavioural Difficulties. 2020 Jan 2;25(1):29-41.
- [Background] Nash P, Renelli M, Stillar A, Streich B, Lafrance A. Long-term outcomes of a brief emotion-focused family therapy intervention for eating disorders across the lifespan: a mixed-methods study. Canadian Journal of Counselling and Psychotherapy. 2020 Apr 14;54(2):130-49.
- [Background] Bode AA, George MW, Weist MD, Stephan SH, Lever N, Youngstrom EA. The impact of parent empowerment in children's mental health services on parenting stress. Journal of Child and Family Studies. 2016 Oct;25(10):3044-55.
- [Background] Gratz KL, Roemer L. Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of psychopathology and behavioral assessment. 2004 Mar;26(1):41-54.
- [Background] Fabes RA, Poulin RE, Eisenberg N, Madden-Derdich DA. The Coping with Children's Negative Emotions Scale (CCNES): Psychometric properties and relations with children's emotional competence. Marriage & Family Review. 2002.
- [Background] Hamilton VE, Matthews JM, Crawford SB. Development and preliminary validation of a parenting self-regulation scale:"me as a parent". Journal of child and family studies. 2015 Oct;24(10):2853-64.
- [Background] Berry JO, Jones WH. The Parental Stress Scale: Initial psychometric evidence. Journal of Social and Personal Relationships. 1995; 12(3), 463-472.
- [Background] Hawley K, Weersing V, Weisz J. The parent and youth consumer satisfaction scales; unpublished questionnaire; 1998.
- [Background] Epstein NB, Baldwin LM, Bishop DS. The McMaster Family Assessment Device. Journal of Marital and Family Therapy. 1983; 9(2), 171-180.
- [Derived] Seddon JA, Reaume CL, Thomassin K. A six-week group program of emotion focused family therapy for parents of children with mental health challenges: protocol for a randomized controlled trial. BMC Psychiatry. 2025 Feb 14;25(1):131. doi: 10.1186/s12888-024-06382-y. PMID 39953468